CLINICAL TRIAL: NCT04129996
Title: Camrelizumab in Combination With Nab-paclitaxel and Famitinib as a First-line Treatment in Patients With Unresectable Locally Advanced or Metastatic Immunomodulatory Triple Negative Breast Cancer: An Open, Single-arm, Multicenter, Efficacy and Safety Phase II Clinical Study.
Brief Title: A Trial of Camrelizumab in Combination With Nab-paclitaxel and Famitinib as a First Line Treatment in Patients With Unresectable Locally Advanced or Metastatic Immunomodulatory Triple Negative Breast Cancer(FUTURE-C-PLUS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, clinical professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N025
Record Dates: First submitted 2019-10-11; First posted 2019-10-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; 130-nm albumin-bound paclitaxel; famitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab in combination with nab-paclitaxel and famitinib (Experimental)
  Interventions: Drug: camrelizumab in combination with nab-paclitaxel and famitinib

INTERVENTIONS:
Drug: camrelizumab in combination with nab-paclitaxel and famitinib — camrelizumab in combination with nab-paclitaxel and famitinib for triple negative breast cancer

SUMMARY:
The study is being conducted to evaluate the efficacy, safety of camrelizumab in combination with nab-paclitaxel and famitinib in Patients with unresectable locally advanced or metastatic immunomodulatory triple negative breast Cancer..

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1
* Expected lifetime of not less than three months
* Metastatic or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression)
* Cancer stage: recurrent or metastatic breast cancer; Local recurrence be confirmed by the researchers could not be radical resection.
* Adequate hematologic and end-organ function, laboratory test results.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1)
* Patients had received no previous chemotherapy or targeted therapy for metastatic triple-negative breast cancer

Exclusion Criteria:

* Previous received anti-VEGFR small molecule tyrosine kinase inhibitors (e.g. famitinib, sorafenib, Sunitinib, regorafenib, etc.) for treatment of the patients .
* A history of bleeding, any serious bleeding events.
* Important blood vessels around tumors has been infringed and high risk of bleeding.
* Coagulant function abnormality
* artery/venous thromboembolism event
* History of autoimmune disease
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Uncontrolled pleural effusion and ascites
* Known central nervous system (CNS) disease.
* Long-term unhealing wound or incomplete healing of fracture
* urine protein ≥2+ and 24h urine protein quantitative > 1 g.
* Pregnancy or lactation.
* Thyroid dysfunction.
* Peripheral neuropathy grade ≥2.
* People with high blood pressure;
* A history of unstable angina;
* New diagnosis of angina pectoris.
* Myocardial infarction incident ;
* Arrhythmia for long-term use of anti-arrhythmic drugs and New York heart association class II or higher cardiac insufficiency

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
ORR | Baseline up to 53 months (assessed at Screening, every 8 weeks for the first 12 months, thereafter every 12 weeks until disease progression or death, whichever occurs first
  Percentage of Participants With an Objective Response of Complete Response (CR) or Partial Response (PR) According to RECIST v1.1 in all Participants

CONTACTS AND LOCATIONS:
Overall Officials: zhimin shao, MD,PHD, Principal Investigator — Fudan University
Locations (1):
- Zhi-Ming Shao, Shanghai, China

REFERENCES:
- [Derived] Wu SY, Xu Y, Chen L, Fan L, Ma XY, Zhao S, Song XQ, Hu X, Yang WT, Chai WJ, Guo XM, Chen XZ, Xu YH, Zhu XY, Zou JJ, Wang ZH, Jiang YZ, Shao ZM. Combined angiogenesis and PD-1 inhibition for immunomodulatory TNBC: concept exploration and biomarker analysis in the FUTURE-C-Plus trial. Mol Cancer. 2022 Mar 25;21(1):84. doi: 10.1186/s12943-022-01536-6. PMID 35337339
- [Derived] Chen L, Jiang YZ, Wu SY, Wu J, Di GH, Liu GY, Yu KD, Fan L, Li JJ, Hou YF, Hu Z, Chen CM, Huang XY, Cao AY, Hu X, Zhao S, Ma XY, Xu Y, Sun XJ, Chai WJ, Guo X, Chen X, Xu Y, Zhu XY, Zou JJ, Yang WT, Wang ZH, Shao ZM. Famitinib with Camrelizumab and Nab-Paclitaxel for Advanced Immunomodulatory Triple-Negative Breast Cancer (FUTURE-C-Plus): An Open-Label, Single-Arm, Phase II Trial. Clin Cancer Res. 2022 Jul 1;28(13):2807-2817. doi: 10.1158/1078-0432.CCR-21-4313. PMID 35247906